CLINICAL TRIAL: NCT03864042
Title: An Open-label Phase 1 Study to Evaluate Drug-Drug Interactions of Agents Co-Administered With Encorafenib and Binimetinib in Patients With BRAF V600-mutant Unresectable or Metastatic Melanoma or Other Advanced Solid Tumors
Brief Title: Pharmacokinetic Drug-drug Interaction Study of Encorafenib and Binimetinib on Probe Drugs in Patients With BRAF V600-mutant Melanoma or Other Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-818-103; C4221003 (Other: Alias Study Number); 2019-001036-66 (EudraCT Number)
Record Dates: First submitted 2019-02-01; First posted 2019-03-06 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors; Metastatic Melanoma
Keywords: solid tumor; melanoma
MeSH Terms: conditions — Melanoma | interventions — Losartan; Dextromethorphan; Caffeine; Omeprazole; Midazolam; Rosuvastatin Calcium; Bupropion; encorafenib; binimetinib; Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 - CYP Probe Cocktail (Experimental): Patients will receive a single oral dose of the CYP Probe Cocktail on Day -7, Day 1, and Day 14:
  * 25 mg losartan oral tablet
  * 30 mg dextromethorphan oral capsule
  * 50 mg caffeine oral liquid
  * 20 mg omeprazole oral capsule
  * 2 mg midazolam oral syrup
  encorafenib/binimetinib continuous daily dosing starting Day 1:
  * 450 mg (6 x 75 mg) encorafenib oral capsules once daily (QD)
  * 45 mg (3 x 15 mg) binimetinib oral tablet twice daily (BID)
  All drugs will be taken within 10 minutes.
  Interventions: Drug: losartan; Drug: dextromethorphan; Drug: caffeine; Drug: omeprazole; Drug: midazolam; Drug: encorafenib; Drug: binimetinib
- Arm 2 - Rosuvastatin and Bupropion (Experimental): Patients will receive a single oral dose of rosuvastatin and bupropion once on Day -7, Day 1 and Day 14:
  * 10 mg rosuvastatin oral tablet
  * 75 mg bupropion immediate release (IR) oral tablet
  encorafenib/binimetinib continuous daily dosing starting Day 1:
  * 450 mg (6 x 75 mg) encorafenib oral capsules once daily (QD)
  * 45 mg (3 x 15 mg) binimetinib oral tablet twice daily (BID)
  All drugs will be taken within 10 minutes.
  Interventions: Drug: rosuvastatin; Drug: bupropion immediate release (IR); Drug: encorafenib; Drug: binimetinib
- Arm 3 - Modafinil (Experimental): Patients will begin encorafenib/binimetinib continuous daily dosing starting Day 1:
  * 450 mg (6 x 75 mg) encorafenib oral capsules once daily (QD)
  * 45 mg (3 x 15 mg) binimetinib oral tablet twice daily (BID)
  then receive continuous treatment of modafinil on Day 15 through Day 21:
  - 400 mg modafinil tablet once daily (QD)
  Interventions: Drug: encorafenib; Drug: binimetinib; Drug: modafinil

INTERVENTIONS:
Drug: losartan — taken orally
  Arms: Arm 1 - CYP Probe Cocktail
Drug: dextromethorphan — taken orally
  Arms: Arm 1 - CYP Probe Cocktail
Drug: caffeine — taken orally
  Arms: Arm 1 - CYP Probe Cocktail
Drug: omeprazole — taken orally
  Arms: Arm 1 - CYP Probe Cocktail
Drug: midazolam — taken orally
  Arms: Arm 1 - CYP Probe Cocktail
Drug: rosuvastatin — taken orally
  Arms: Arm 2 - Rosuvastatin and Bupropion
Drug: bupropion immediate release (IR) — taken orally
  Arms: Arm 2 - Rosuvastatin and Bupropion
Drug: encorafenib — taken orally
Drug: binimetinib — taken orally
Drug: modafinil — taken orally
  Arms: Arm 3 - Modafinil

SUMMARY:
This is an open-label, 3-arm, fixed-sequence study to evaluate the effect of single and multiple oral doses of encorafenib in combination with binimetinib on the single oral dose pharmacokinetics (PK) of cytochrome P450 (CYP) enzyme probe substrates using a probe cocktail, on an organic anion-transporting polypeptide/breast cancer resistance protein (OATP/BCRP) substrate using rosuvastatin and on a CYP2B6 substrate using bupropion. The effect of multiple oral doses of the moderate cytochrome P450 (CYP) inhibitor modafinil on encorafenib in combination with binimetinib will also be assessed. The study will have 2 treatment phases, a drug-drug interaction (DDI) phase followed by a post-DDI phase.

ELIGIBILITY:
Key Inclusion Criteria - Patients must meet all of the inclusion criteria to be eligible for enrollment into the study:

* Histologically confirmed diagnosis of locally advanced, unresectable or metastatic cutaneous melanoma or unknown primary melanoma American Joint Committee on Cancer (AJCC) Stage IIIB, IIIC or IV; or other BRAF V600-mutant advanced solid tumors
* Presence of BRAF V600E and/or V600K mutation in tumor tissue prior to enrollment, as determined using a local test;
* Evidence of measurable or non-measurable lesions
* Patient with unresectable locally advanced or metastatic melanoma who has received no prior treatment or progressed on or after prior systemic therapy; Note: Prior therapy with a BRAF proto-oncogene serine-threonine protein kinase (BRAF) inhibitor and/or a mitogen-activated protein (MAP) kinase (MEK) inhibitor is permitted except in the regimen immediately prior to study entry
* Patient with other (non-melanoma) BRAF V600E and/or V600K -mutant advanced solid tumors who has progressed on standard therapy or for whom there are no available standard therapies; Note: Prior therapy with a BRAF inhibitor and/or a MEK inhibitor is permitted except in the regimen immediately prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Adequate bone marrow, hepatic and renal function as specified in the protocol
* ARM 1 ONLY: Non-smoker who has not used nicotine containing products for at least 3 months prior to the first dose.

Key Exclusion Criteria - Patients meeting any of the following criteria are not eligible for enrollment in the study:

* Symptomatic brain metastasis. Patients previously treated or untreated for these conditions that are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Brain metastases must be stable, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT] demonstrating no current evidence of progressive brain metastases at screening);
* Symptomatic or untreated leptomeningeal disease;
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes);
* Clinically significant cardiac disease
* Known hyper-coagulability risks other than malignancy (e.g., Factor V Leiden syndrome);
* Thromboembolic event except catheter-related venous thrombosis ≤ 12 weeks prior to starting study treatment.
* Discontinuation of prior BRAF and/or MEK inhibitor treatment due to left ventricular dysfunction, pneumonitis/interstitial lung disease, or retinal vein occlusion;
* ARM 1 ONLY: Positive urine cotinine test at screening
* ARM 3 ONLY:

  * History of psychosis, depression or mania;
  * History of angioedema;
  * History of mitral valve prolapse;
  * History of left ventricular hypertrophy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2023-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (11):
  - UC Irvine Health, Orange, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Illinois at Chicago, Chicago, Illinois
  - Hopkins Eye Clinic, Hopkins, Minnesota
  - Park Nicollet Eye Clinic, Maple Grove, Minnesota
  - Regions Cancer Care Center, Saint Paul, Minnesota
  - HealthPartners Specialty Center-Eye Care, Saint Paul, Minnesota
  - Gabrail Cancer Center Research, Canton, Ohio
  - University of TN Medical Center, Knoxville, Tennessee
  - Mary Crowley Cancer Research - Medical City Hospital, Dallas, Texas
  - Utah Cancer Specialists, West Valley City, Utah
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Jewish General Hospital, Montrea, Quebec
- Netherlands (2):
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - Erasmus Medical Center, Rotterdam
- Spain (10):
  - Hospital del Mar, Barcelona
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Beata Maria Ana, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Rementeria, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - CERCO, Seville
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Piscitelli J, Reddy MB, Wollenberg L, Del Frari L, Gong J, Matschke K, Williams JH. Evaluation of the effect of modafinil on the pharmacokinetics of encorafenib and binimetinib in patients with BRAF V600-mutant advanced solid tumors. Cancer Chemother Pharmacol. 2024 Sep;94(3):337-347. doi: 10.1007/s00280-024-04676-2. Epub 2024 Jun 15. PMID 38878209
- [Derived] Piscitelli J, Reddy MB, Wollenberg L, Del Frari L, Gong J, Wood L, Zhang Y, Matschke K, Williams JH. Clinical Evaluation of the Effect of Encorafenib on Bupropion, Rosuvastatin, and Coproporphyrin I and Considerations for Statin Coadministration. Clin Pharmacokinet. 2024 Apr;63(4):483-496. doi: 10.1007/s40262-024-01352-9. Epub 2024 Feb 29. PMID 38424308
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=ARRAY-818-103

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in 3 Arms to evaluate the potential drug-drug interactions (DDIs) of single and multiple oral doses of encorafenib in combination with binimetinib with sensitive substrates of specific cytochrome P450 (CYP) enzymes (Arm 1), organic anion-transporting polypeptide (OATP)/breast cancer resistance protein (BCRP) transporters (Arm 2), and moderate CYP3A4 inducer (Arm 3). A total of 29, 12, 15 participants were enrolled in Arm 1, Arm 2, and Arm 3, respectively.
Groups:
- Arm 1 - CYP Probe Cocktail: Participants received a single oral dose of the CYP probe cocktail (losartan tablet 25 milligrams [mg], dextromethorphan capsule 30 mg, caffeine liquid 50 mg, omeprazole capsule 20 mg, and midazolam syrup 2 mg) on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg once daily [QD]) and binimetinib (tablet, 45 mg twice daily [BID]) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
- Arm 2 - Rosuvastatin and Bupropion: Participants received a single oral dose of rosuvastatin tablet 10 mg and bupropion immediate release (IR) tablet 75 mg on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
- Arm 3 - Modafinil: Participants received continuous treatment with encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) from Day 1 until treatment discontinuation criteria were met. Continuous treatment of modafinil (tablet, 400 mg QD) was started on Day 15 through Day 21. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 28 days (Day 1 to Day 28).
Period: DDI Phase
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion | Arm 3 - Modafinil
Started | 29 | 12 | 15
Completed | 25 | 12 | 15
Not Completed | 4 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0
Period: Post-DDI Phase
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion | Arm 3 - Modafinil
Started | 25 | 12 | 15
Completed | 0 | 0 | 0
Not Completed | 25 | 12 | 15
Not completed — Adverse Event | 5 | 3 | 2
Not completed — Progressive Disease | 11 | 6 | 13
Not completed — Discretion of investigator | 1 | 1 | 0
Not completed — Study terminated by sponsor | 7 | 0 | 0
Not completed — Withdrawal of consent | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population who were treated with encorafenib-binimetinib.
Groups:
- Arm 1 - CYP Probe Cocktail: Participants received a single oral dose of the CYP probe cocktail (losartan tablet 25 mg, dextromethorphan capsule 30 mg, caffeine liquid 50 mg, omeprazole capsule 20 mg, and midazolam syrup 2 mg) on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
- Arm 2 - Rosuvastatin and Bupropion: Participants received a single oral dose of rosuvastatin tablet 10 mg and bupropion IR tablet 75 mg on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
- Arm 3 - Modafinil: Participants received continuous treatment with encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) from Day 1 until treatment discontinuation criteria were met.continuous treatment of modafinil (tablet, 400 mg QD) was started on Day 15 through Day 21. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 28 days (Day 1 to Day 28).
- Total: Total of all reporting groups
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion | Arm 3 - Modafinil | Total
Number analyzed (Participants) | 27 | 12 | 15 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (12.14) | 61.3 (13.65) | 58.9 (9.98) | 61.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 7 | 27
  Male | 13 | 6 | 8 | 27
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 25 | 11 | 14 | 50
  Black or African American | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 2
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Plasma Midazolam on Day -7, Day 1, and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: All participants in Arm 1 who received at least 1 dose of any study intervention and had at least 1 post-baseline pharmacokinetic (PK) sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Days -7, 1, and 14. Number of participants analyzed represents the total number of participants in Arm 1 in the evaluable PK set. Number analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
nanograms per milliliter (ng/mL)
  Day -7 | 9.45 (45.1)
  Day 1 | 11.1 (50.6)
  Day 14 | 2.44 (54.6)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.17, 90% CI 2-sided [0.978 to 1.40] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.258, 90% CI 2-sided [0.215 to 0.308] — Day 14 / Day -7

2. Primary Outcome: Cmax of Plasma Total 1-OH Midazolam on Day -7, Day 1, and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data. The metabolites of midazolam included total 1-OH midazolam, free 1-OH midazolam, and glucuronide conjugated 1-hydroxymidazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: All participants in Arm 1 who received at least 1 dose of any study intervention and had at least 1 post-baseline PK sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Days -7, 1, and 14. Number of participants analyzed represents the total number of participants in Arm 1 in the evaluable PK set. Number analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng/mL
  Day -7 | 45.2 (31.5)
  Day 1 | 50.5 (40.8)
  Day 14 | 56.7 (27.7)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.12, 90% CI 2-sided [0.998 to 1.25] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.25, 90% CI 2-sided [1.12 to 1.40] — Day 14 / Day -7

3. Primary Outcome: Cmax of Plasma Free 1-OH Midazolam on Day -7, Day 1, and Day 14
Description: as for outcome 2
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng/mL
  Day -7 | 3.36 (53.4)
  Day 1 | 4.52 (52.7)
  Day 14 | 2.09 (71.6)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.34, 90% CI 2-sided [1.12 to 1.62] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.622, 90% CI 2-sided [0.517 to 0.748] — Day 14 / Day -7

4. Primary Outcome: Cmax of Plasma Glucuronide Conjugated 1-Hydroxymidazolam on Day -7, Day 1, and Day 14
Description: as for outcome 2
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng/mL
  Day -7 | 41.5 (32.8)
  Day 1 | 45.4 (43.7)
  Day 14 | 54.1 (29.1)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.09, 90% CI 2-sided [0.975 to 1.23] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.30, 90% CI 2-sided [1.16 to 1.46] — Day 14 / Day -7

5. Primary Outcome: Cmax of Plasma Absolute Caffeine on Day -7, Day 1, and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data. Due to dietary caffeine intake may resulted in positive pre-dose concentrations, absolute and/or baseline-adjusted caffeine were analyzed. Baseline adjusted concentration = measured concentration - [predose concentration*e^(-Kel*t)], where Kel is terminal elimination rate constant based on actual measured concentration values for each profile and t is the actual sampling time.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng/mL
  Day -7: number analyzed (Participants) | 15
  Day -7 | 1150 (31.5)
  Day 1: number analyzed (Participants) | 15
  Day 1 | 1210 (30.6)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 1300 (19.8)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.05, 90% CI 2-sided [0.922 to 1.20] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.13, 90% CI 2-sided [0.992 to 1.29] — Day 14 / Day -7

6. Primary Outcome: Cmax of Plasma Baseline-Adjusted Caffeine on Day -7, Day 1, and Day 14
Description: as for outcome 5
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng/mL
  Day -7: number analyzed (Participants) | 18
  Day -7 | 984 (37.2)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 1070 (40.4)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 1110 (29.7)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.09, 90% CI 2-sided [0.990 to 1.19] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.10, 90% CI 2-sided [1.00 to 1.22] — Day 14 / Day -7

7. Primary Outcome: Cmax of Plasma Paraxanthine on Day -7, Day 1, and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data. Paraxanthine was the metabolite of caffeine.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng/mL
  Day -7: number analyzed (Participants) | 15
  Day -7 | 357 (41.6)
  Day 1: number analyzed (Participants) | 15
  Day 1 | 319 (27.7)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 247 (53.5)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.894, 90% CI 2-sided [0.741 to 1.08] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.692, 90% CI 2-sided [0.573 to 0.835] — Day 14 / Day -7

8. Primary Outcome: Cmax of Plasma Omeprazole on Day -7, Day 1, and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng/mL
  Day -7 | 267 (188.7)
  Day 1 | 354 (73.1)
  Day 14 | 271 (57.1)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.32, 90% CI 2-sided [0.861 to 2.04] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.01, 90% CI 2-sided [0.659 to 1.56] — Day 14 / Day -7

9. Primary Outcome: Cmax of Plasma 5-OH Omeprazole on Day -7, Day 1, and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng/mL
  Day -7 | 91.8 (104.5)
  Day 1 | 90.4 (79.3)
  Day 14 | 64.4 (54.8)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.01, 90% CI 2-sided [0.762 to 1.33] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.718, 90% CI 2-sided [0.543 to 0.948] — Day 14 / Day -7

10. Primary Outcome: Cmax of Plasma Rosuvastatin on Day -7, Day 1 and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: All participants in Arm 2 who received at least 1 dose of any study intervention and had at least 1 post-baseline PK sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Days -7, 1, and 14. Number of participants analyzed represents the total number of participants in Arm 2 in the evaluable PK set. Number analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Arm 2 - Rosuvastatin and Bupropion: Participants received a single oral dose of rosuvastatin tablet 10 mg and bupropion IR tablet 75 mg on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All drugs were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
ng/mL
  Day -7 | 6.98 (96.4)
  Day 1 | 30.3 (130.8)
  Day 14 | 18.7 (113.7)
Statistical Analysis 1: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 4.34, 90% CI 2-sided [2.94 to 6.40] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 2.68, 90% CI 2-sided [1.82 to 3.96] — Day 14 / Day -7

11. Primary Outcome: Cmax of Plasma Bupropion on Day -7, Day 1 and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
ng/mL
  Day -7 | 94.0 (63.9)
  Day 1 | 70.9 (50.6)
  Day 14 | 71.0 (52.7)
Statistical Analysis 1: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 0.754, 90% CI 2-sided [0.595 to 0.954] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 0.755, 90% CI 2-sided [0.596 to 0.957] — Day 14 / Day -7

12. Primary Outcome: Cmax of Plasma Hydroxybupropion on Day -7, Day 1 and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data. Hydroxybupropion was the metabolite of bupropion.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
ng/mL
  Day -7 | 181 (46.9)
  Day 1 | 189 (49.7)
  Day 14 | 256 (62.5)
Statistical Analysis 1: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 1.05, 90% CI 2-sided [0.864 to 1.27] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 1.42, 90% CI 2-sided [1.17 to 1.72] — Day 14 / Day -7

13. Primary Outcome: Area Under the Concentration-Time Profile From Time 0 to The Time of The Last Quantifiable Concentration (AUClast) of Plasma Midazolam on Day -7, Day 1, and Day 14
Description: AUClast is area under the concentration-time profile (AUC) from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
nanograms*hour per milliliter (ng*hr/mL)
  Day -7 | 25.7 (57.2)
  Day 1 | 27.6 (58.4)
  Day 14 | 4.52 (52.9)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.07, 90% CI 2-sided [0.920 to 1.25] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.175, 90% CI 2-sided [0.151 to 0.204] — Day 14 / Day -7

14. Primary Outcome: AUClast of Plasma Total 1-OH Midazolam on Day -7, Day 1, and Day 14
Description: AUClast is AUC from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method. The metabolites of midazolam included total 1-OH midazolam, free 1-OH midazolam, and glucuronide conjugated 1-hydroxymidazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7 | 135 (29.9)
  Day 1 | 173 (41.8)
  Day 14 | 142 (38.9)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.28, 90% CI 2-sided [1.18 to 1.38] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.05, 90% CI 2-sided [0.974 to 1.14] — Day 14 / Day -7

15. Primary Outcome: AUClast of Plasma Free 1-OH Midazolam on Day -7, Day 1, and Day 14
Description: as for outcome 14
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7 | 8.87 (43.7)
  Day 1 | 11.1 (46.6)
  Day 14 | 4.55 (62.6)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.25, 90% CI 2-sided [1.09 to 1.43] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.513, 90% CI 2-sided [0.449 to 0.587] — Day 14 / Day -7

16. Primary Outcome: AUClast of Plasma Glucuronide Conjugated 1-Hydroxymidazolam on Day -7, Day 1, and Day 14
Description: as for outcome 14
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7 | 125 (32.0)
  Day 1 | 160 (44.5)
  Day 14 | 133 (41.0)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.28, 90% CI 2-sided [1.17 to 1.39] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.07, 90% CI 2-sided [0.979 to 1.16] — Day 14 / Day -7

17. Primary Outcome: AUClast of Plasma Absolute Caffeine on Day -7, Day 1, and Day 14
Description: AUClast is AUC from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method. Due to dietary caffeine intake may resulted in positive pre-dose concentrations, absolute and/or baseline-adjusted caffeine were analyzed. Baseline adjusted concentration = measured concentration - [predose concentration*e^(-Kel*t)], where Kel is terminal elimination rate constant based on actual measured concentration values for each profile and t is the actual sampling time.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 15
  Day -7 | 5940 (35.8)
  Day 1: number analyzed (Participants) | 15
  Day 1 | 6480 (34.4)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 7520 (22.7)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.09, 90% CI 2-sided [0.947 to 1.26] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.27, 90% CI 2-sided [1.10 to 1.46] — Day 14 / Day -7

18. Primary Outcome: AUClast of Plasma Baseline-Adjusted Caffeine on Day -7, Day 1, and Day 14
Description: as for outcome 17
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 18
  Day -7 | 5100 (36.6)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 5700 (45.7)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 6430 (29.6)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.12, 90% CI 2-sided [1.02 to 1.23] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.26, 90% CI 2-sided [1.14 to 1.38] — Day 14 / Day -7

19. Primary Outcome: AUClast of Plasma Paraxanthine on Day -7, Day 1, and Day 14
Description: AUClast is AUC from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method. Paraxanthine was the metabolite of caffeine.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 15
  Day -7 | 2160 (47.7)
  Day 1: number analyzed (Participants) | 15
  Day 1 | 1940 (31.5)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 1470 (64.6)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.900, 90% CI 2-sided [0.721 to 1.12] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.679, 90% CI 2-sided [0.544 to 0.848] — Day 14 / Day -7

20. Primary Outcome: AUClast of Plasma Omeprazole on Day -7, Day 1, and Day 14
Description: AUClast is AUC from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7 | 815 (193.3)
  Day 1 | 1020 (91.9)
  Day 14 | 674 (54.3)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.26, 90% CI 2-sided [0.800 to 1.98] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.827, 90% CI 2-sided [0.526 to 1.30] — Day 14 / Day -7

21. Primary Outcome: AUClast of Plasma 5-OH Omeprazole in Arm 1 on Day -7, Day 1 and Day 14
Description: AUClast is AUC from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 18
  Day -7 | 313 (134.6)
  Day 1 | 302 (92.1)
  Day 14 | 195 (60.6)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.980, 90% CI 2-sided [0.688 to 1.39] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.633, 90% CI 2-sided [0.445 to 0.900] — Day 14 / Day -7

22. Primary Outcome: AUClast of Plasma Rosuvastatin on Day -7, Day 1 and Day 14
Description: as for outcome 20
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
ng*hr/mL
  Day -7 | 33.6 (88.1)
  Day 1 | 93.8 (97.9)
  Day 14 | 52.8 (66.3)
Statistical Analysis 1: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 2.79, 90% CI 2-sided [2.08 to 3.74] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 1.57, 90% CI 2-sided [1.17 to 2.11] — Day 14 / Day -7

23. Primary Outcome: AUClast of Plasma Bupropion on Day -7, Day 1 and Day 14
Description: as for outcome 20
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
ng*hr/mL
  Day -7 | 339 (48.1)
  Day 1 | 261 (49.0)
  Day 14 | 250 (50.1)
Statistical Analysis 1: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 0.769, 90% CI 2-sided [0.637 to 0.928] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 0.736, 90% CI 2-sided [0.610 to 0.889] — Day 14 / Day -7

24. Primary Outcome: AUClast of Plasma Hydroxybupropion on Day -7, Day 1 and Day 14
Description: AUClast is AUC from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method. Hydroxybupropion was the metabolite of bupropion.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
ng*hr/mL
  Day -7 | 1090 (59.8)
  Day 1 | 1080 (63.8)
  Day 14 | 1610 (65.7)
Statistical Analysis 1: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 0.993, 90% CI 2-sided [0.803 to 1.23] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 2 - Rosuvastatin and Bupropion; Test type: Other; Geometric LS Mean Ratio = 1.48, 90% CI 2-sided [1.20 to 1.83] — Day 14 / Day -7

25. Primary Outcome: The Amount Eliminated Via Urine Over an 8-Hour Period (Ae0-8) of Losartan on Day -7, Day 1 and Day 14
Description: Ae0-8 is the amount excreted into the urine over the collection interval of 0 to 8 hours.
Time Frame: 0 to 8 hours after dosing on Days -7, 1 and 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams (mg)
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
milligrams (mg)
  Day -7: number analyzed (Participants) | 17
  Day -7 | 0.239 (268.0)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.349 (314.2)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 0.286 (277.3)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.45, 90% CI 2-sided [0.902 to 2.32] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.18, 90% CI 2-sided [0.720 to 1.93] — Day 14 / Day -7

26. Primary Outcome: Ae0-8 of E-3174 on Day -7, Day 1 and Day 14
Description: Ae0-8 is the amount excreted into the urine over the collection interval of 0 to 8 hours. E-3174 was the metabolite of losartan.
Time Frame: 0 to 8 hours after dosing on Days -7, 1 and 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
mg
  Day -7: number analyzed (Participants) | 17
  Day -7 | 0.227 (293.3)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.332 (276.2)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 0.205 (317.8)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.47, 90% CI 2-sided [0.915 to 2.36] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.851, 90% CI 2-sided [0.519 to 1.39] — Day 14 / Day -7

27. Primary Outcome: Ae0-8 of Dextromethorphan on Day -7, Day 1 and Day 14
Description: Ae0-8 is the amount excreted into the urine over the collection interval of 0 to 8 hours.
Time Frame: 0 to 8 hours after dosing on Days -7, 1 and 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
mg
  Day -7: number analyzed (Participants) | 17
  Day -7 | 0.0264 (396.7)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.0323 (542.5)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 0.0225 (899.2)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.20, 90% CI 2-sided [0.775 to 1.87] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.940, 90% CI 2-sided [0.593 to 1.49] — Day 14 / Day -7

28. Primary Outcome: Ae0-8 of Dextrorphan on Day -7, Day 1 and Day 14
Description: Ae0-8 is the amount excreted into the urine over the collection interval of 0 to 8 hours. Dextrorphan was the metabolite of dextromethorphan.
Time Frame: 0 to 8 hours after dosing on Days -7, 1 and 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
mg
  Day -7: number analyzed (Participants) | 17
  Day -7 | 3.78 (183.9)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 4.41 (165.5)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 3.55 (222.5)
Statistical Analysis 1: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 1.18, 90% CI 2-sided [0.830 to 1.67] — Day 1 / Day -7
Statistical Analysis 2: Comparison: Arm 1 - CYP Probe Cocktail; Test type: Other; Geometric LS Mean Ratio = 0.979, 90% CI 2-sided [0.680 to 1.41] — Day 14 / Day -7

29. Primary Outcome: Cmax of Plasma Encorafenib on Day 14 and Day 21 in Arm 3
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: All participants in Arm 3 who received at least 1 dose of any study intervention and had at least 1 post-baseline PK sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Days 14 and 21. Number of participants analyzed represents the total number of participants in Arm 3 in the evaluable PK set. Number analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Arm 3 - Modafinil: Participants received continuous treatment with encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) from Day 1 until treatment discontinuation criteria were met. Continuous treatment of modafinil (tablet, 400 mg QD) was started on Day 15 through Day 21. All drugs were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 28 days (Day 1 to Day 28).
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
ng/mL
  Day 14 | 3540 (55.6)
  Day 21 | 2830 (67.2)
Statistical Analysis 1: Comparison: Arm 3 - Modafinil; Test type: Other; Geometric LS Mean Ratio = 0.798, 90% CI 2-sided [0.585 to 1.09] — Day 21 / Day 14

30. Primary Outcome: Cmax of Plasma LHY746 on Day 14 and Day 21 in Arm 3
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data. LHY746 was the metabolite of encorafenib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
ng/mL
  Day 14 | 2460 (24.7)
  Day 21 | 2510 (26.8)
Statistical Analysis 1: Comparison: Arm 3 - Modafinil; Test type: Other; Geometric LS Mean Ratio = 1.02, 90% CI 2-sided [0.935 to 1.11] — Day 21 / Day 14

31. Primary Outcome: AUClast of Plasma Encorafenib on Day 14 and Day 21 in Arm 3
Description: as for outcome 20
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
ng*hr/mL
  Day 14 | 11900 (35.8)
  Day 21 | 9100 (30.3)
Statistical Analysis 1: Comparison: Arm 3 - Modafinil; Test type: Other; Geometric LS Mean Ratio = 0.762, 90% CI 2-sided [0.613 to 0.945] — Day 21 / Day 14

32. Primary Outcome: AUClast of Plasma LHY746 on Day 14 and Day 21 in Arm 3
Description: AUClast is AUC from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method. LHY746 was the metabolite of encorafenib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
ng*hr/mL
  Day 14 | 31100 (45.4)
  Day 21 | 33100 (31.2)
Statistical Analysis 1: Comparison: Arm 3 - Modafinil; Test type: Other; Geometric LS Mean Ratio = 1.06, 90% CI 2-sided [0.929 to 1.22] — Day 21 / Day 14

33. Secondary Outcome: Ratio of AUClast Values of the Metabolite Compared to Parent (MRAUClast) for 1-OH Midazolam/Midazolam on Day -7, Day 1 and Day 14
Description: MRAUClast is the ratio of AUClast values of the metabolite compared to parent, corrected for molecular weight (MW), which was calculated by [AUClast (metabolite) × MW (parent)] / [AUClast (parent) × MW (metabolite)]. 1-OH midazolam was the metabolite of midazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7 | 5.00 (63.3)
  Day 1 | 5.97 (72.6)
  Day 14 | 30.1 (65.7)

34. Secondary Outcome: Ratio of AUC From Time Zero Extrapolated to Infinity (AUCinf) Values of the Metabolite Compared to Parent (MRAUCinf) for 1-OH Midazolam/Midazolam on Day -7, Day 1 and Day 14
Description: MRAUCinf is the ratio of AUCinf values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [AUCinf (metabolite) × MW (parent)] / [AUCinf (parent) × MW (metabolite)]. 1-OH midazolam was the metabolite of midazolam. AUCinf is AUC from time zero to extrapolated infinite time. It is obtained by AUClast + (Clast/kel), where AUClast is the AUC from time zero to the time of last quantifiable concentration (Clast), and kel is the apparent terminal elimination rate constant.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7: number analyzed (Participants) | 16
  Day -7 | 4.31 (68.6)
  Day 1: number analyzed (Participants) | 8
  Day 1 | 5.21 (87.8)
  Day 14: number analyzed (Participants) | 14
  Day 14 | 29.5 (70.3)

35. Secondary Outcome: MRAUClast for Paraxanthine/Caffeine on Day -7, Day 1 and Day 14
Description: MRAUClast is the ratio of AUClast values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [AUClast (metabolite) × MW (parent)] / [AUClast (parent) × MW (metabolite)]. Paraxanthine was the metabolite of caffeine.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7: number analyzed (Participants) | 15
  Day -7 | 0.392 (37.2)
  Day 1: number analyzed (Participants) | 15
  Day 1 | 0.324 (44.5)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 0.211 (72.3)

36. Secondary Outcome: MRAUClast for 5-OH Omeprazole/Omeprazole on Day -7, Day 1 and Day 14
Description: MRAUClast is the ratio of AUClast values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [AUClast (metabolite) × MW (parent)] / [AUClast (parent) × MW (metabolite)]. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7: number analyzed (Participants) | 18
  Day -7 | 0.309 (107.2)
  Day 1 | 0.282 (87.0)
  Day 14 | 0.277 (44.6)

37. Secondary Outcome: MRAUCinf for 5-OH Omeprazole/Omeprazole on Day -7, Day 1 and Day 14
Description: MRAUCinf is the ratio of AUCinf values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [AUCinf (metabolite) × MW (parent)] / [AUCinf (parent) × MW (metabolite)]. 5-OH Omeprazole was the metabolite of omeprazole. AUCinf is AUC from time zero to extrapolated infinite time. It is obtained by AUClast + (Clast/kel), where AUClast is the AUC from time zero to the time of last quantifiable concentration (Clast), and kel is the apparent terminal elimination rate constant.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 18
Ratio
  Day -7: number analyzed (Participants) | 5
  Day -7 | 0.312 (119.8)
  Day 1: number analyzed (Participants) | 2
  Day 1 | 0.960 (92.6)
  Day 14: number analyzed (Participants) | 11
  Day 14 | 0.312 (49.8)

38. Secondary Outcome: MRAUClast for Hydroxybupropion/Bupropion on Day -7, Day 1 and Day 14
Description: MRAUClast is the ratio of AUClast values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [AUClast (metabolite) × MW (parent)] / [AUClast (parent) × MW (metabolite)]. Hydroxybupropion was the metabolite of bupropion.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
Ratio
  Day -7 | 3.01 (60.2)
  Day 1 | 3.88 (47.5)
  Day 14 | 6.04 (57.5)

39. Secondary Outcome: MRAUClast for LHY746/Encorafenib in Arm 3 on Day 14 and Day 21
Description: MRAUClast is the ratio of AUClast values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [AUClast (metabolite) × MW (parent)] / [AUClast (parent) × MW (metabolite)]. LHY746 was the metabolite of encorafenib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Ratio
  Day 14 | 3.31 (58.9)
  Day 21 | 4.62 (43.3)

40. Secondary Outcome: Ratio of Cmax Values of the Metabolite Compared to Parent (MRCmax) for 1-OH Midazolam/Midazolam on Day -7, Day 1 and Day 14
Description: MRCmax is the ratio of Cmax values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [Cmax (metabolite) × MW (parent)] / [Cmax (parent) × MW (metabolite)]. 1-OH midazolam was the metabolite of midazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7 | 4.56 (54.7)
  Day 1 | 4.36 (62.8)
  Day 14 | 22.2 (60.6)

41. Secondary Outcome: MRCmax for Paraxanthine/Caffeine on Day -7, Day 1 and Day 14
Description: MRCmax is the ratio of Cmax values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [Cmax (metabolite) × MW (parent)] / [Cmax (parent) × MW (metabolite)]. Paraxanthine was the metabolite of caffeine.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7: number analyzed (Participants) | 15
  Day -7 | 0.335 (25.4)
  Day 1: number analyzed (Participants) | 15
  Day 1 | 0.285 (36.8)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 0.205 (54.9)

42. Secondary Outcome: MRCmax for 5-OH Omeprazole/Omeprazole on Day -7, Day 1 and Day 14
Description: MRCmax is the ratio of Cmax values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [Cmax (metabolite) × MW (parent)] / [Cmax (parent) × MW (metabolite)]. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7 | 0.273 (115.2)
  Day 1 | 0.244 (83.0)
  Day 14 | 0.227 (48.2)

43. Secondary Outcome: MRCmax for Hydroxybupropion/Bupropion on Day -7, Day 1 and Day 14
Description: MRCmax is the ratio of Cmax values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [Cmax (metabolite) × MW (parent)] / [Cmax (parent) × MW (metabolite)]. Hydroxybupropion was the metabolite of bupropion.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
Ratio
  Day -7 | 1.80 (61.1)
  Day 1 | 2.51 (50.0)
  Day 14 | 3.38 (48.8)

44. Secondary Outcome: MRCmax for LHY746/Encorafenib in Arm 3 on Day 14 and Day 21
Description: MRCmax is the ratio of Cmax values of the metabolite compared to parent, corrected for molecular weight, which was calculated by [Cmax (metabolite) × MW (parent)] / [Cmax (parent) × MW (metabolite)]. LHY746 was the metabolite of encorafenib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Ratio
  Day 14 | 0.883 (72.5)
  Day 21 | 1.13 (77.6)

45. Secondary Outcome: Ratio of Ae0-8 Values of the Metabolite Compared to Parent (MRAe0-8) for E-3174/Losartan on Day -7, Day 1 and Day 14
Description: Ae0-8 is the amount excreted into the urine over the collection interval of 0 to 8 hours. MRAe0-8 is the ratio of Ae0-8 values of the metabolite compared to parent, corrected for molecular weight. E-3174 was the metabolite of losartan.
Time Frame: 0 to 8 hours after dosing on Days -7, 1 and 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7: number analyzed (Participants) | 17
  Day -7 | 0.920 (65.6)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.921 (100.0)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 0.693 (99.0)

46. Secondary Outcome: MRAe0-8 for Dextrorphan/Dextromethorphan on Day -7, Day 1 and Day 14
Description: Ae0-8 is the amount excreted into the urine over the collection interval of 0 to 8 hours. MRAe0-8 is the ratio of Ae0-8 values of the metabolite compared to parent, corrected for molecular weight. Dextrorphan was the metabolite of dextromethorphan.
Time Frame: 0 to 8 hours after dosing on Days -7, 1 and 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Ratio
  Day -7: number analyzed (Participants) | 17
  Day -7 | 151 (383.2)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 144 (560.9)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 167 (354.5)

47. Secondary Outcome: Time to Reach Cmax (Tmax) of Plasma Midazolam on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 1.00 [0.77 to 2.93]
  Day 1 | 0.88 [0.77 to 1.30]
  Day 14 | 0.88 [0.68 to 1.00]

48. Secondary Outcome: Tmax of Plasma Total 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data. The metabolites of midazolam included total 1-OH midazolam, free 1-OH midazolam, and glucuronide conjugated 1-hydroxymidazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14.
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 1.00 [0.77 to 2.93]
  Day 1 | 0.90 [0.80 to 1.85]
  Day 14 | 0.88 [0.68 to 1.00]

49. Secondary Outcome: Tmax of Plasma Free 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: as for outcome 48
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 1.00 [0.77 to 2.93]
  Day 1 | 0.90 [0.80 to 1.85]
  Day 14 | 0.92 [0.68 to 1.72]

50. Secondary Outcome: Tmax of Plasma Glucuronide Conjugated 1-Hydroxymidazolam on Day -7, Day 1 and Day 14
Description: as for outcome 48
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 1.00 [0.77 to 2.97]
  Day 1 | 0.90 [0.80 to 1.83]
  Day 14 | 0.88 [0.68 to 1.00]

51. Secondary Outcome: Tmax of Plasma Absolute Caffeine on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data. Due to dietary caffeine intake may resulted in positive pre-dose concentrations, absolute and/or baseline-adjusted caffeine were analyzed. Baseline adjusted concentration = measured concentration - [predose concentration*e^(-Kel*t)], where Kel is terminal elimination rate constant based on actual measured concentration values for each profile and t is the actual sampling time.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7: number analyzed (Participants) | 15
  Day -7 | 1.00 [0.80 to 1.98]
  Day 1: number analyzed (Participants) | 15
  Day 1 | 0.93 [0.78 to 1.88]
  Day 14: number analyzed (Participants) | 15
  Day 14 | 0.90 [0.72 to 2.92]

52. Secondary Outcome: Tmax of Plasma Baseline-Adjusted Caffeine on Day -7, Day 1 and Day 14
Description: as for outcome 51
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7: number analyzed (Participants) | 18
  Day -7 | 1.00 [0.80 to 2.17]
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.94 [0.78 to 1.88]
  Day 14: number analyzed (Participants) | 17
  Day 14 | 0.98 [0.72 to 3.97]

53. Secondary Outcome: Tmax of Plasma Paraxanthine on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data. Paraxanthine was the metabolite of caffeine.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7: number analyzed (Participants) | 15
  Day -7 | 7.18 [3.77 to 7.98]
  Day 1: number analyzed (Participants) | 15
  Day 1 | 7.63 [1.83 to 7.92]
  Day 14: number analyzed (Participants) | 15
  Day 14 | 6.00 [2.13 to 8.00]

54. Secondary Outcome: Tmax of Plasma Omeprazole on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours (+/- 15 minutes window for each time-point) postdose on Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 2.20 [1.05 to 8.07]
  Day 1 | 3.00 [0.87 to 7.92]
  Day 14 | 3.00 [0.85 to 7.85]

55. Secondary Outcome: Tmax of Plasma 5-OH Omeprazole on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours (+/- 15 minutes window for each time-point) postdose on Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 2.97 [0.00 to 8.07]
  Day 1 | 3.80 [0.87 to 7.92]
  Day 14 | 3.00 [0.85 to 7.85]

56. Secondary Outcome: Tmax of Plasma Rosuvastatin on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
Hours
  Day -7 | 2.40 [1.00 to 4.02]
  Day 1 | 1.85 [0.78 to 7.00]
  Day 14 | 1.40 [0.92 to 3.00]

57. Secondary Outcome: Tmax of Plasma Bupropion on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
Hours
  Day -7 | 1.87 [0.82 to 4.00]
  Day 1 | 1.93 [0.77 to 4.00]
  Day 14 | 1.92 [0.93 to 2.87]

58. Secondary Outcome: Tmax of Plasma Hydroxybupropion on Day -7, Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data. Hydroxybupropion was the metabolite of bupropion.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
Hours
  Day -7 | 4.00 [3.00 to 8.00]
  Day 1 | 7.68 [3.83 to 8.00]
  Day 14 | 3.94 [1.00 to 6.17]

59. Secondary Outcome: AUCinf of Plasma Midazolam on Day -7, Day 1 and Day 14
Description: AUCinf is AUC from time zero to extrapolated infinite time. It is obtained by AUClast + (Clast/kel), where AUClast is the AUC from time zero to the time of last quantifiable concentration (Clast), and kel is the apparent terminal elimination rate constant.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 9
  Day -7 | 27.1 (72.5)
  Day 1: number analyzed (Participants) | 10
  Day 1 | 27.1 (65.1)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 5.10 (52.5)

60. Secondary Outcome: AUCinf of Plasma Total 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: AUCinf is AUC from time zero to extrapolated infinite time. It is obtained by AUClast + (Clast/kel), where AUClast is the AUC from time zero to the time of last quantifiable concentration (Clast), and kel is the apparent terminal elimination rate constant. The metabolites of midazolam included total 1-OH midazolam, free 1-OH midazolam, and glucuronide conjugated 1-hydroxymidazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 16
  Day -7 | 150 (27.7)
  Day 1: number analyzed (Participants) | 8
  Day 1 | 172 (49.1)
  Day 14: number analyzed (Participants) | 14
  Day 14 | 154 (35.5)

61. Secondary Outcome: AUCinf of Plasma Free 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: as for outcome 60
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 15
  Day -7 | 9.98 (43.9)
  Day 1: number analyzed (Participants) | 17
  Day 1 | 13.1 (44.9)
  Day 14: number analyzed (Participants) | 14
  Day 14 | 5.52 (56.2)

62. Secondary Outcome: AUCinf of Plasma Glucuronide Conjugated 1-Hydroxymidazolam on Day -7, Day 1 and Day 14
Description: as for outcome 60
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 15
  Day -7 | 139 (30.6)
  Day 1: number analyzed (Participants) | 7
  Day 1 | 167 (52.4)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 143 (36.3)

63. Secondary Outcome: AUCinf of Plasma Omeprazole on Day -7, Day 1 and Day 14
Description: as for outcome 59
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
ng*hr/mL
  Day -7: number analyzed (Participants) | 8
  Day -7 | 1630 (151.6)
  Day 1: number analyzed (Participants) | 5
  Day 1 | 1170 (79.4)
  Day 14: number analyzed (Participants) | 12
  Day 14 | 904 (35.7)

64. Secondary Outcome: AUCinf of Plasma 5-OH Omeprazole on Day -7, Day 1 and Day 14
Description: AUCinf is AUC from time zero to extrapolated infinite time. It is obtained by AUClast + (Clast/kel), where AUClast is the AUC from time zero to the time of last quantifiable concentration (Clast), and kel is the apparent terminal elimination rate constant. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 18
ng*hr/mL
  Day -7: number analyzed (Participants) | 5
  Day -7 | 557 (92.6)
  Day 1: number analyzed (Participants) | 2
  Day 1 | 880 (21.8)
  Day 14: number analyzed (Participants) | 11
  Day 14 | 294 (44.5)

65. Secondary Outcome: AUCinf of Plasma Rosuvastatin on Day -7, Day 1 and Day 14
Description: as for outcome 59
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
ng*hr/mL
  Day -7: number analyzed (Participants) | 2
  Day -7 | 75.4 (62.3)
  Day 1: number analyzed (Participants) | 7
  Day 1 | 139 (69.8)
  Day 14: number analyzed (Participants) | 8
  Day 14 | 62.9 (48.5)

66. Secondary Outcome: AUCinf of Plasma Bupropion on Day -7, Day 1 and Day 14
Description: as for outcome 59
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
ng*hr/mL
  Day -7: number analyzed (Participants) | 6
  Day -7 | 398 (54.9)
  Day 1: number analyzed (Participants) | 2
  Day 1 | 390 (11.1)
  Day 14: number analyzed (Participants) | 8
  Day 14 | 298 (38.4)

67. Secondary Outcome: Percent of AUC Extrapolated (AUC%Extrap) of Plasma Midazolam on Day -7, Day 1 and Day 14
Description: AUC%extrap is the percentage of AUCinf obtained by forward extrapolation. It is calculated as (AUCinf minus AUClast)*100/ AUCinf.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
percentage of AUC
  Day -7 | 19.1 (46.0)
  Day 1 | 19.3 (37.6)
  Day 14 | 8.76 (55.2)

68. Secondary Outcome: AUC%Extrap of Plasma Total 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: AUC%extrap is the percentage of AUCinf obtained by forward extrapolation. It is calculated as (AUCinf minus AUClast)*100/ AUCinf. The metabolites of midazolam included total 1-OH midazolam, free 1-OH midazolam, and glucuronide conjugated 1-hydroxymidazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of AUC
  Day -7 | 15.2 (35.2)
  Day 1 | 21.9 (40.1)
  Day 14 | 12.6 (68.4)

69. Secondary Outcome: AUC%Extrap of Plasma Free 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: as for outcome 68
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of AUC
  Day -7 | 14.1 (42.6)
  Day 1 | 12.9 (46.1)
  Day 14 | 12.8 (68.1)

70. Secondary Outcome: AUC%Extrap of Plasma Glucuronide Conjugated 1-Hydroxymidazolam on Day -7, Day 1 and Day 14
Description: as for outcome 68
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of AUC
  Day -7: number analyzed (Participants) | 18
  Day -7 | 15.3 (35.0)
  Day 1 | 22.6 (40.5)
  Day 14 | 14.1 (54.9)

71. Secondary Outcome: AUC%Extrap of Plasma Absolute Caffeine on Day -7, Day 1 and Day 14
Description: AUC%extrap is the percentage of AUCinf obtained by forward extrapolation. It is calculated as (AUCinf minus AUClast)*100/ AUCinf. Due to dietary caffeine intake may resulted in positive pre-dose concentrations, absolute and/or baseline-adjusted caffeine were analyzed. Baseline adjusted concentration = measured concentration - [predose concentration*e^(-Kel*t)], where Kel is terminal elimination rate constant based on actual measured concentration values for each profile and t is the actual sampling time.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of AUC
  Day -7: number analyzed (Participants) | 14
  Day -7 | 48.3 (39.4)
  Day 1: number analyzed (Participants) | 14
  Day 1 | 53.2 (27.0)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 61.0 (26.0)

72. Secondary Outcome: AUC%Extrap of Plasma Baseline-Adjusted Caffeine on Day -7, Day 1 and Day 14
Description: as for outcome 71
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of AUC
  Day -7: number analyzed (Participants) | 16
  Day -7 | 46.7 (37.6)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 54.8 (25.5)
  Day 14: number analyzed (Participants) | 13
  Day 14 | 58.0 (25.3)

73. Secondary Outcome: AUC%Extrap of Plasma Omeprazole on Day -7, Day 1 and Day 14
Description: as for outcome 67
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of AUC
  Day -7: number analyzed (Participants) | 9
  Day -7 | 7.35 (142.1)
  Day 1: number analyzed (Participants) | 8
  Day 1 | 11.9 (141.2)
  Day 14: number analyzed (Participants) | 13
  Day 14 | 4.22 (113.9)

74. Secondary Outcome: AUC%Extrap of Plasma 5-OH Omeprazole on Day -7, Day 1 and Day 14
Description: AUC%extrap is the percentage of AUCinf obtained by forward extrapolation. It is calculated as (AUCinf minus AUClast)*100/ AUCinf. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of AUC
  Day -7: number analyzed (Participants) | 7
  Day -7 | 12.4 (147.3)
  Day 1: number analyzed (Participants) | 9
  Day 1 | 26.1 (65.7)
  Day 14: number analyzed (Participants) | 12
  Day 14 | 8.07 (66.7)

75. Secondary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Plasma Midazolam on Day -7, Day 1 and Day 14
Description: Kel is the apparent terminal elimination rate constant, which is estimated by linear regression of time versus loge concentration.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour
  Day -7 | 0.196 (26.2)
  Day 1 | 0.188 (22.6)
  Day 14 | 0.347 (55.4)

76. Secondary Outcome: Kel of Plasma Total 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: Kel is the apparent terminal elimination rate constant, which is estimated by linear regression of time versus loge concentration. The metabolites of midazolam included total 1-OH midazolam, free 1-OH midazolam, and glucuronide conjugated 1-hydroxymidazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour
  Day -7 | 0.248 (20.1)
  Day 1 | 0.199 (31.3)
  Day 14 | 0.259 (36.9)

77. Secondary Outcome: Kel of Plasma Free 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: as for outcome 76
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour
  Day -7 | 0.231 (24.2)
  Day 1 | 0.236 (31.1)
  Day 14 | 0.269 (47.2)

78. Secondary Outcome: Kel of Plasma Glucuronide Conjugated 1-Hydroxymidazolam on Day -7, Day 1 and Day 14
Description: as for outcome 76
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour
  Day -7: number analyzed (Participants) | 18
  Day -7 | 0.241 (23.3)
  Day 1 | 0.197 (32.5)
  Day 14 | 0.277 (37.7)

79. Secondary Outcome: Kel of Plasma Absolute Caffeine on Day -7, Day 1 and Day 14
Description: Kel is the apparent terminal elimination rate constant, which is estimated by linear regression of time versus loge concentration. Due to dietary caffeine intake may resulted in positive pre-dose concentrations, absolute and/or baseline-adjusted caffeine were analyzed. Baseline adjusted concentration = measured concentration - [predose concentration*e^(-Kel*t)], where Kel is terminal elimination rate constant based on actual measured concentration values for each profile and t is the actual sampling time.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour
  Day -7: number analyzed (Participants) | 14
  Day -7 | 0.0870 (57.4)
  Day 1: number analyzed (Participants) | 14
  Day 1 | 0.0753 (61.3)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 0.0575 (61.7)

80. Secondary Outcome: Kel of Plasma Baseline-Adjusted Caffeine on Day -7, Day 1 and Day 14
Description: as for outcome 79
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour
  Day -7: number analyzed (Participants) | 16
  Day -7 | 0.0893 (70.3)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.0739 (58.3)
  Day 14: number analyzed (Participants) | 13
  Day 14 | 0.0656 (54.4)

81. Secondary Outcome: Kel of Plasma Omeprazole on Day -7, Day 1 and Day 14
Description: as for outcome 75
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour
  Day -7: number analyzed (Participants) | 9
  Day -7 | 0.401 (50.4)
  Day 1: number analyzed (Participants) | 8
  Day 1 | 0.296 (53.1)
  Day 14: number analyzed (Participants) | 13
  Day 14 | 0.461 (31.1)

82. Secondary Outcome: Kel of Plasma 5-OH Omeprazole on Day -7, Day 1 and Day 14
Description: Kel is the apparent terminal elimination rate constant, which is estimated by linear regression of time versus loge concentration. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour
  Day -7: number analyzed (Participants) | 7
  Day -7 | 0.303 (43.1)
  Day 1: number analyzed (Participants) | 9
  Day 1 | 0.197 (45.7)
  Day 14: number analyzed (Participants) | 12
  Day 14 | 0.386 (22.5)

83. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of Plasma Midazolam on Day -7, Day 1 and Day 14
Description: T1/2 is the terminal elimination half-life, which is estimated by Loge(2) / kel, where kel is the apparent terminal elimination rate constant.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 3.54 (26.2)
  Day 1 | 3.69 (22.6)
  Day 14 | 2.00 (55.4)

84. Secondary Outcome: T1/2 of Plasma Total 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: T1/2 is the terminal elimination half-life, which is estimated by Loge(2) / kel, where kel is the apparent terminal elimination rate constant. The metabolites of midazolam included total 1-OH midazolam, free 1-OH midazolam, and glucuronide conjugated 1-hydroxymidazolam.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 2.80 (20.1)
  Day 1 | 3.48 (31.3)
  Day 14 | 2.68 (36.9)

85. Secondary Outcome: T1/2 of Plasma Free 1-OH Midazolam on Day -7, Day 1 and Day 14
Description: as for outcome 84
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7 | 3.00 (24.2)
  Day 1 | 2.93 (31.1)
  Day 14 | 2.58 (47.2)

86. Secondary Outcome: T1/2 of Plasma Glucuronide Conjugated 1-Hydroxymidazolam on Day -7, Day 1 and Day 14
Description: as for outcome 84
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7: number analyzed (Participants) | 18
  Day -7 | 2.87 (23.3)
  Day 1 | 3.53 (32.5)
  Day 14 | 2.50 (37.7)

87. Secondary Outcome: T1/2 of Plasma Absolute Caffeine on Day -7, Day 1 and Day 14
Description: T1/2 is the terminal elimination half-life, which is estimated by Loge(2) / kel, where kel is the apparent terminal elimination rate constant. Due to dietary caffeine intake may resulted in positive pre-dose concentrations, absolute and/or baseline-adjusted caffeine were analyzed. Baseline adjusted concentration = measured concentration - [predose concentration*e^(-Kel*t)], where Kel is terminal elimination rate constant based on actual measured concentration values for each profile and t is the actual sampling time.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7: number analyzed (Participants) | 14
  Day -7 | 7.97 (57.4)
  Day 1: number analyzed (Participants) | 14
  Day 1 | 9.20 (61.3)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 12.1 (61.7)

88. Secondary Outcome: T1/2 of Plasma Baseline-Adjusted Caffeine on Day -7, Day 1 and Day 14
Description: as for outcome 87
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7: number analyzed (Participants) | 16
  Day -7 | 7.76 (70.3)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 9.38 (58.3)
  Day 14: number analyzed (Participants) | 13
  Day 14 | 10.6 (54.4)

89. Secondary Outcome: T1/2 of Plasma Omeprazole on Day -7, Day 1 and Day 14
Description: as for outcome 83
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7: number analyzed (Participants) | 9
  Day -7 | 1.73 (50.4)
  Day 1: number analyzed (Participants) | 8
  Day 1 | 2.34 (53.1)
  Day 14: number analyzed (Participants) | 13
  Day 14 | 1.50 (31.1)

90. Secondary Outcome: T1/2 of Plasma 5-OH Omeprazole on Day -7, Day 1 and Day 14
Description: T1/2 is the terminal elimination half-life, which is estimated by Loge(2) / kel, where kel is the apparent terminal elimination rate constant. 5-OH Omeprazole was the metabolite of omeprazole.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Hours
  Day -7: number analyzed (Participants) | 7
  Day -7 | 2.29 (43.1)
  Day 1: number analyzed (Participants) | 9
  Day 1 | 3.53 (45.7)
  Day 14: number analyzed (Participants) | 12
  Day 14 | 1.80 (22.5)

91. Secondary Outcome: T1/2 of Plasma Rosuvastatin on Day -7, Day 1 and Day 14
Description: as for outcome 83
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
Hours
  Day -7: number analyzed (Participants) | 5
  Day -7 | 3.25 (51.8)
  Day 1: number analyzed (Participants) | 7
  Day 1 | 2.13 (17.0)
  Day 14: number analyzed (Participants) | 8
  Day 14 | 1.86 (23.0)

92. Secondary Outcome: T1/2 of Plasma Bupropion on Day -7, Day 1 and Day 14
Description: as for outcome 83
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 10
Hours
  Day -7: number analyzed (Participants) | 7
  Day -7 | 2.81 (15.1)
  Day 1: number analyzed (Participants) | 7
  Day 1 | 3.24 (10.2)
  Day 14: number analyzed (Participants) | 9
  Day 14 | 2.75 (15.2)

93. Secondary Outcome: Apparent Clearance (CL/F) of Plasma Midazolam on Day -7, Day 1 and Day 14
Description: CL/F is the apparent total body clearance of drug from the plasma (parent drugs only), which is estimated by Dose / AUCinf (Day -7) or Dose / AUClast (Day 1 and Day 14).
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)/hour (h)
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Liters (L)/hour (h)
  Day -7: number analyzed (Participants) | 9
  Day -7 | 73.9 (72.5)
  Day 1: number analyzed (Participants) | 10
  Day 1 | 73.9 (65.1)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 392 (52.5)

94. Secondary Outcome: CL/F of Plasma Omeprazole on Day -7, Day 1 and Day 14
Description: as for outcome 93
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
L/h
  Day -7: number analyzed (Participants) | 8
  Day -7 | 12.3 (151.6)
  Day 1: number analyzed (Participants) | 5
  Day 1 | 17.0 (79.4)
  Day 14: number analyzed (Participants) | 12
  Day 14 | 22.1 (35.7)

95. Secondary Outcome: Apparent Total Volume of Distribution Following Oral Administration (Vz/F) of Plasma Midazolam on Day -7, Day 1 and Day 14
Description: Vz/F is the apparent volume of distribution during the terminal phase (parent drugs only), which is calculated by CL/F/kel.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Litre
  Day -7: number analyzed (Participants) | 9
  Day -7 | 306 (67.7)
  Day 1: number analyzed (Participants) | 10
  Day 1 | 339 (54.6)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 1030 (54.7)

96. Secondary Outcome: Vz/F of Plasma Omeprazole on Day -7, Day 1 and Day 14
Description: as for outcome 95
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Litre
  Day -7: number analyzed (Participants) | 8
  Day -7 | 29.1 (93.9)
  Day 1: number analyzed (Participants) | 5
  Day 1 | 44.6 (63.7)
  Day 14: number analyzed (Participants) | 12
  Day 14 | 45.9 (39.3)

97. Secondary Outcome: Percentage of Dose Recovered in Urine (Fe) for Losartan on Day -7, Day 1 and Day 14
Description: Fe is the percentage of dose recovered in urine from 0 to 8 hours as parent or metabolite, which was calculated as Ae0-8 / dose × 100.
Time Frame: Predose, and 0 to 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of dose
  Day -7: number analyzed (Participants) | 17
  Day -7 | 0.478 (268.0)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.699 (314.2)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 0.572 (277.3)

98. Secondary Outcome: Fe for E-3174 on Day -7, Day 1 and Day 14
Description: Fe is the percentage of dose recovered in urine from 0 to 8 hours as parent or metabolite, which was calculated as Ae0-8 / dose × 100. E-3174 was the metabolite of losartan.
Time Frame: 0 to 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of dose
  Day -7: number analyzed (Participants) | 17
  Day -7 | 0.440 (293.3)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.644 (276.2)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 0.396 (317.8)

99. Secondary Outcome: Fe for Dextromethorphan on Day -7, Day 1 and Day 14
Description: as for outcome 97
Time Frame: 0 to 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of dose
  Day -7: number analyzed (Participants) | 17
  Day -7 | 0.0881 (396.7)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 0.108 (542.5)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 0.0750 (899.2)

100. Secondary Outcome: Fe for Dextrorphan on Day -7, Day 1 and Day 14
Description: Fe is the percentage of dose recovered in urine from 0 to 8 hours as parent or metabolite, which was calculated as Ae0-8 / dose × 100. Dextrorphan was the metabolite of dextromethorphan.
Time Frame: 0 to 8 hours postdose on Day -7, Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of dose
  Day -7: number analyzed (Participants) | 17
  Day -7 | 13.3 (183.9)
  Day 1: number analyzed (Participants) | 18
  Day 1 | 15.6 (165.5)
  Day 14: number analyzed (Participants) | 17
  Day 14 | 12.5 (222.5)

101. Secondary Outcome: Cmax of Encorafenib on Day 1 and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14.
Population: All participants in Arms 1 and 2 who received at least 1 dose of any study intervention and had at least 1 post-baseline PK sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Days 1 and 14. Number of participants analyzed represents the total number of participants in each arm in the evaluable PK set. Number analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
ng/mL
  Day 1 | 6150 (41.9) | 6060 (77.7)
  Day 14 | 3240 (55.7) | 2940 (72.2)

102. Secondary Outcome: Cmax of LHY746 on Day 1 and Day 14
Description: as for outcome 30
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
ng/mL
  Day 1 | 943 (66.6) | 953 (66.0)
  Day 14 | 2490 (32.4) | 2340 (66.8)

103. Secondary Outcome: Cmax of Binimetinib on Day 1 and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14.
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
ng/mL
  Day 1 | 661 (55.1) | 549 (89.5)
  Day 14 | 521 (59.9) | 566 (63.1)

104. Secondary Outcome: Cmax of AR00426032 on Day 1 and Day 14
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data. AR00426032 was the metabolite of binimetinib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
ng/mL
  Day 1 | 57.0 (41.2) | 63.3 (73.2)
  Day 14 | 23.3 (85.6) | 27.4 (43.1)

105. Secondary Outcome: AUClast of Encorafenib on Day 1 and Day 14
Description: as for outcome 20
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14.
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
ng*hr/mL
  Day 1 | 24500 (36.7) | 25900 (61.7)
  Day 14 | 12700 (37.6) | 13100 (28.6)

106. Secondary Outcome: AUClast of LHY746 on Day 1 and Day 14
Description: as for outcome 32
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
ng*hr/mL
  Day 1 | 5130 (66.1) | 4990 (78.1)
  Day 14 | 34000 (34.4) | 32800 (54.5)

107. Secondary Outcome: AUClast of Binimetinib on Day 1 and Day 14
Description: as for outcome 20
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
ng*hr/mL
  Day 1 | 2290 (43.3) | 2040 (81.0)
  Day 14 | 2190 (33.8) | 2210 (40.7)

108. Secondary Outcome: AUClast of AR00426032 on Day 1 and Day 14
Description: AUClast is AUC from time 0 to the time of the last quantifiable concentration. It was calculated using the linear trapezoidal/linear interpolation method. AR00426032 was the metabolite of binimetinib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
ng*hr/mL
  Day 1 | 236 (39.6) | 256 (74.8)
  Day 14 | 108 (74.1) | 122 (67.4)

109. Secondary Outcome: Tmax of Encorafenib on Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14.
Population: as for outcome 101
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
Hours
  Day 1 | 2.00 [1.00 to 5.92] | 1.87 [0.85 to 3.98]
  Day 14 | 1.94 [0.82 to 3.02] | 1.93 [1.00 to 4.00]

110. Secondary Outcome: Tmax of LHY746 on Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data. LHY746 was the metabolite of encorafenib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours (+/- 15 minutes window for each time-point) postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
Hours
  Day 1 | 6.93 [2.07 to 8.07] | 7.42 [3.00 to 8.00]
  Day 14 | 2.98 [1.80 to 8.22] | 3.47 [1.85 to 6.25]

111. Secondary Outcome: Tmax of Binimetinib on Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14.
Population: as for outcome 101
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
Hours
  Day 1 | 1.97 [0.87 to 4.03] | 1.97 [0.85 to 4.08]
  Day 14 | 1.98 [0.97 to 3.02] | 1.93 [1.02 to 2.92]

112. Secondary Outcome: Tmax of AR00426032 on Day 1 and Day 14
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data. AR00426032 was the metabolite of binimetinib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
Hours
  Day 1 | 2.02 [0.98 to 4.03] | 2.48 [1.82 to 6.13]
  Day 14 | 2.00 [0.98 to 3.02] | 2.00 [1.00 to 2.92]

113. Secondary Outcome: AUCinf of Encorafenib on Day 1
Description: as for outcome 59
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: All participants in Arms 1 and 2 who received at least 1 dose of any study intervention and had at least 1 post-baseline PK sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Day 1. Number of participants analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 4 | 3
ng*hr/mL | 26200 (71.6) | 45100 (56.8)

114. Secondary Outcome: AUCinf of Binimetinib on Day 1
Description: as for outcome 59
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1.
Population: as for outcome 113
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 12 | 6
ng*hr/mL | 2970 (45.4) | 3280 (47.7)

115. Secondary Outcome: AUCinf of AR00426032 on Day 1
Description: as for outcome 59
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: All participants in Arms 1 and 2 who received at least 1 dose of any study intervention and had at least 1 post-baseline PK sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Day 1. Number of participants analyzed represents the total number of participants in each arm in the evaluable PK set. Number of analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 9 | 2
ng*hr/mL | 270 (40.5) | 432 (32.4)

116. Secondary Outcome: T1/2 of Encorafenib on Day 1 and Day 14
Description: as for outcome 83
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
Hours
  Day 1: number analyzed (Participants) | 19 | 7
  Day 1 | 3.98 (46.4) | 3.77 (37.0)
  Day 14 | 4.37 (42.7) | 3.58 (13.7)

117. Secondary Outcome: T1/2 of LHY746 on Day 1 and Day 14
Description: T1/2 is the terminal elimination half-life, which is estimated by Loge(2) / kel, where kel is the apparent terminal elimination rate constant. LHY746 was the metabolite of encorafenib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
Hours
  Day 1: number analyzed (Participants) | 2 | 1
  Day 1 | 9.47 (130.1) | 22.5 (NA) — Data was not reported as only 1 participant was analyzed for this arm.
  Day 14: number analyzed (Participants) | 19 | 6
  Day 14 | 9.27 (40.0) | 11.2 (20.6)

118. Secondary Outcome: T1/2 of Binimetinib on Day 1 and Day 14
Description: as for outcome 83
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
Hours
  Day 1: number analyzed (Participants) | 17 | 6
  Day 1 | 2.62 (35.4) | 2.45 (17.3)
  Day 14: number analyzed (Participants) | 19 | 10
  Day 14 | 3.90 (39.9) | 3.70 (42.8)

119. Secondary Outcome: T1/2 of AR00426032 on Day 1 and Day 14
Description: T1/2 is the terminal elimination half-life, which is estimated by Loge(2) / kel, where kel is the apparent terminal elimination rate constant. AR00426032 was the metabolite of binimetinib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1 and Day 14
Population: as for outcome 101
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion
Number analyzed (Participants) | 20 | 10
Hours
  Day 1: number analyzed (Participants) | 17 | 6
  Day 1 | 2.96 (23.3) | 3.15 (24.7)
  Day 14: number analyzed (Participants) | 16 | 9
  Day 14 | 3.97 (42.6) | 3.89 (51.9)

120. Secondary Outcome: AUC%Extrap of Encorafenib on Day 1
Description: as for outcome 67
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: All participants in Arm 1 who received at least 1 dose of any study intervention and had at least 1 post-baseline PK sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Day 1. Number of participants analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Percentage of AUC | 24.4 (73.9)

121. Secondary Outcome: AUC%Extrap of LHY746 on Day 1
Description: AUC%extrap is the percentage of AUCinf obtained by forward extrapolation. It is calculated as (AUCinf minus AUClast)*100/ AUCinf. LHY746 was the metabolite of encorafenib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 2
Percentage of AUC | 52.9 (56.1)

122. Secondary Outcome: AUC%Extrap of Binimetinib on Day 1
Description: as for outcome 67
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 17
Percentage of AUC | 13.7 (60.2)

123. Secondary Outcome: AUC%Extrap of AR00426032 on Day 1
Description: AUC%extrap is the percentage of AUCinf obtained by forward extrapolation. It is calculated as (AUCinf minus AUClast)*100/ AUCinf. AR00426032 was the metabolite of binimetinib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 17
Percentage of AUC | 19.8 (33.8)

124. Secondary Outcome: Kel of Encorafenib on Day 1
Description: as for outcome 75
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 19
Fraction/hour | 0.174 (46.4)

125. Secondary Outcome: Kel of LHY746 on Day 1
Description: Kel is the apparent terminal elimination rate constant, which is estimated by linear regression of time versus loge concentration. LHY746 was the metabolite of encorafenib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 2
Fraction/hour | 0.0732 (130.1)

126. Secondary Outcome: Kel of Binimetinib on Day 1
Description: as for outcome 75
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 17
Fraction/hour | 0.265 (35.4)

127. Secondary Outcome: Kel of AR00426032 on Day 1
Description: Kel is the apparent terminal elimination rate constant, which is estimated by linear regression of time versus loge concentration. AR00426032 was the metabolite of binimetinib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction/hour
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 17
Fraction/hour | 0.234 (23.3)

128. Secondary Outcome: CL/F of Encorafenib on Day 1
Description: as for outcome 93
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1.
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 4
L/h | 17.2 (71.6)

129. Secondary Outcome: CL/F of Binimetinib on Day 1
Description: as for outcome 93
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1.
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 12
L/h | 15.1 (45.4)

130. Secondary Outcome: Vz/F of Encorafenib on Day 1
Description: as for outcome 95
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1.
Population: All participants in Arm 1 who received at least 1 dose of any study intervention and had at least 1 post-baseline PK sample with an associated bioanalytical result, and who were with sufficient concentration data to calculate at least 1 PK parameter on Day 1. Number of participants analyzed represents the total number of participants in Arm 1 in the evaluable PK set. Number of analyzed represents the number of participants who had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 4
Litre | 53.4 (38.2)

131. Secondary Outcome: Vz/F of Binimetinib on Day 1
Description: as for outcome 95
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 1.
Population: as for outcome 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Arm 1 - CYP Probe Cocktail
Number analyzed (Participants) | 12
Litre | 47.6 (50.5)

132. Secondary Outcome: Cmax of Binimetinib on Day 14 and Day 21
Description: Cmax is the maximum plasma concentration which was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
ng/mL
  Day 14 | 660 (39.7)
  Day 21 | 663 (25.3)

133. Secondary Outcome: Cmax of AR00426032 on Day 14 and Day 21
Description: as for outcome 104
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
ng/mL
  Day 14 | 25.9 (63.2)
  Day 21 | 24.7 (36.7)

134. Secondary Outcome: AUClast of Binimetinib on Day 14 and Day 21
Description: as for outcome 20
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
ng*hr/mL
  Day 14 | 2400 (38.6)
  Day 21 | 2290 (30.6)

135. Secondary Outcome: AUClast of AR00426032 on Day 14 and Day 21
Description: AUClast is AUC from time 0 (pre-dose) to the time of the last quantifiable concentration. AR00426032 was the metabolite of binimetinib.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
ng*hr/mL
  Day 14 | 114 (64.5)
  Day 21 | 112 (33.0)

136. Secondary Outcome: Tmax of Encorafenib on Day 14 and Day 21
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Hours
  Day 14 | 1.00 [0.88 to 2.03]
  Day 21 | 1.00 [0.98 to 3.00]

137. Secondary Outcome: Tmax of LHY746 on Day 14 and Day 21
Description: as for outcome 110
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Hours
  Day 14 | 2.05 [1.00 to 6.00]
  Day 21 | 2.10 [1.00 to 6.00]

138. Secondary Outcome: Tmax of Binimetinib on Day 14 and Day 21
Description: Tmax is time to reach maximum observed plasma concentration. It was observed directly from the concentration-time data.
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Hours
  Day 14 | 1.00 [0.88 to 3.00]
  Day 21 | 1.00 [0.95 to 2.10]

139. Secondary Outcome: Tmax of AR00426032 on Day 14 and Day 21
Description: as for outcome 112
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Hours
  Day 14 | 2.00 [0.88 to 3.00]
  Day 21 | 2.00 [0.95 to 2.23]

140. Secondary Outcome: T1/2 of Encorafenib on Day 14 and Day 21
Description: as for outcome 83
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Hours
  Day 14 | 3.48 (26.6)
  Day 21 | 3.57 (27.3)

141. Secondary Outcome: T1/2 of LHY746 on Day 14 and Day 21
Description: as for outcome 117
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Hours
  Day 14: number analyzed (Participants) | 9
  Day 14 | 8.67 (33.1)
  Day 21: number analyzed (Participants) | 10
  Day 21 | 8.01 (18.8)

142. Secondary Outcome: T1/2 of Binimetinib on Day 14 and Day 21
Description: as for outcome 83
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Hours
  Day 14 | 4.62 (42.1)
  Day 21 | 4.55 (44.8)

143. Secondary Outcome: T1/2 of AR00426032 on Day 14 and Day 21
Description: as for outcome 119
Time Frame: Predose, and 1, 2, 3, 4, 6 and 8 hours postdose on Day 14 and Day 21
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Arm 3 - Modafinil
Number analyzed (Participants) | 11
Hours
  Day 14 | 5.60 (37.1)
  Day 21 | 5.22 (58.7)

144. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in the DDI Phase
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were those with initial onset or increasing in severity between the first dose of encorafenib/binimetinib and up to 30 days after treatment discontinuation. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. SAEs were adjudicated according to the investigator's assessment. Treatment-related AEs and SAEs were determined by the investigator.
Time Frame: After 1st dose of encorafenib/binimetinib on Day 1 and up to Day 28 visit in the DDI Phase
Population: All participants who received at least 1 dose of encorafenib/binimetinib.
Measure: Number; unit: Count of Participants
Groups:
- Arm 1 - CYP Probe Cocktail (DDI Phase): Participants received a single oral dose of the CYP probe cocktail (losartan tablet 25 mg, dextromethorphan capsule 30 mg, caffeine liquid 50 mg, omeprazole capsule 20 mg, and midazolam syrup 2 mg) on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All drugs were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
- Arm 2 - Rosuvastatin and Bupropion (DDI Phase): Participants received a single oral dose of rosuvastatin tablet 10 mg and bupropion IR tablet 75 mg on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All drugs were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
- Arm 3 - Modafinil (DDI Phase): Participants received continuous treatment with encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) from Day 1 until treatment discontinuation criteria were met. Continuous treatment of modafinil (tablet, 400 mg QD) was started on Day 15 through Day 21. All drugs were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 28 days (Day 1 to Day 28).
Arm/Group | Arm 1 - CYP Probe Cocktail (DDI Phase) | Arm 2 - Rosuvastatin and Bupropion (DDI Phase) | Arm 3 - Modafinil (DDI Phase)
Number analyzed (Participants) | 27 | 12 | 15
Count of Participants
  Participants with all-causality TEAEs | 26 | 9 | 11
  Participants with treatment-related TEAEs | 24 | 6 | 10
  Participants with all-causality SAEs | 2 | 1 | 0
  Participants with treatment-related SAEs | 1 | 1 | 0
  AEs leading to study drug discontinuation (all-causality) | 3 | 2 | 0
  AEs leading to study drug discontinuation (treatment-related) | 2 | 2 | 0
  AEs requiring dose interruption (all-causality) | 10 | 4 | 4
  AEs requiring dose interruption (treatment-related) | 8 | 2 | 2
  AEs requiring dose reduction (all-causality) | 2 | 2 | 0
  AEs requiring dose reduction (treatment-related) | 2 | 2 | 0
  AEs requiring additional therapy (all-causality) | 13 | 8 | 10
  AEs requiring additional therapy (treatment-related) | 8 | 6 | 8
  Deaths | 0 | 0 | 0

145. Secondary Outcome: Number of Participants With Laboratory Abnormalities in the DDI Phase
Description: Laboratory parameters:hematology (hemoglobin,hematocrit,red blood cell [RBC],platelet,white blood cell count [WBC],neutrophils,eosinophils,monocytes, basophils, lymphocytes), chemistry (albumin, alkaline phosphatase, alanine aminotransferase, amylase, aspartate aminotransferase, bicarbonate, total bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lactate dehydrogenase, lipase, magnesium, inorganic phosphate, potassium, total protein, sodium, uric acid), urinalysis (appearance, color, specific gravity, pH, ketones, protein, glucose, blood, nitrates, leukocyte esterase, and urine microscopy results including WBC, RBC, bacteria, epithelial cells, and casts), coagulation (activated partial thromboplastin time, prothrombin time/international normalized ratio) and others. Clinically notable: worsening from baseline by at least 2 grades or to greater than or equal to (>=) Grade 3, by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.
Time Frame: After 1st dose of encorafenib/binimetinib on Day 1 and up to Day 28 visit in the DDI Phase
Population: All participants who received at least 1 dose of encorafenib/binimetinib.
Measure: Number; unit: Count of Participants
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion | Arm 3 - Modafinil
Number analyzed (Participants) | 27 | 12 | 15
Count of Participants
  Hemoglobin CTCAE Graded Low | 0 | 1 | 0
  Lymphocytes CTCAE Graded Low | 3 | 2 | 0
  Lymphocytes CTCAE Graded High | 2 | 0 | 0
  Neutrophils CTCAE Graded Low | 2 | 1 | 0
  Amylase CTCAE Graded High | 2 | 0 | 1
  Creatinine CTCAE Graded High | 2 | 0 | 3
  Glucose CTCAE Graded High | 2 | 1 | 1
  Lipase CTCAE Graded High | 7 | 0 | 0
  Glucose CTCAE Graded Low | 0 | 1 | 1
  Creatine Kinase CTCAE Graded High | 0 | 2 | 0

146. Secondary Outcome: Number of Participants With Notable Abnormalities in Vital Signs in the DDI Phase
Description: Vital signs (temperature, pulse rate [PR]), systolic blood pressure [SBP]), and diastolic blood pressure [DBP]) were obtained with participants following at least 5 minutes of supine rest. Categorical criteria were defined as DBP>=100 millimeters of mercury (mm Hg)/less than or equal to (<=) 50 mmHg with increase/decrease from baseline of >=15 mmHg; SBP: >=160 mmHg/<=90 mmHg with increase/decrease from baseline of >=20 mmHg; PR: >=120 beats per minute (bpm)/<=50 bpm with increase/decrease from baseline of >=15 bpm; temperature for Arms 1 and 3: >=37.5°C/<=35°C; Arms 2: >=37.5°C/<=36°C.
Time Frame: After 1st dose of encorafenib/binimetinib on Day 1 and up to Day 28 visit in the DDI Phase
Population: All participants who received at least 1 dose of encorafenib/binimetinib.
Measure: Number; unit: Count of Participants
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion | Arm 3 - Modafinil
Number analyzed (Participants) | 27 | 12 | 15
Count of Participants
  SBP high (>=160mmHg with increase from baseline of >=20mmHg) | 4 | 4 | 0
  SBP low (<=90mmHg with decrease from baseline of >=20mmHg) | 0 | 0 | 1
  DBP high (>=100mmHg with increase from baseline of >=15mmHg) | 1 | 0 | 0
  DBP low (<=50mmHg with decrease from baseline of >=15mmHg) | 0 | 0 | 1
  PR high (>=120bpm with increase from baseline of >=15bpm) | 1 | 1 | 0
  PR low (<=50bpm with decrease from baseline of >=15bpm） | 0 | 0 | 1
  Temperature high: number analyzed (Participants) | 27 | 10 | 14
  Temperature high | 0 | 2 | 0
  Temperature low: number analyzed (Participants) | 27 | 10 | 14
  Temperature low | 2 | 3 | 1

147. Secondary Outcome: Number of Participants With Notable Electrocardiogram (ECG) Findings in the DDI Phase
Description: Triplicate 12-lead ECG were performed after the participant had rested quietly for at least 10 minutes in a supine position. ECG parameters included RR interval, PR interval, QRS complex, QT interval, corrected QT (QTc) interval, Bazett's correction QT (QTcB) interval, Heart Rate and Fridericia's correction (QTcF) interval. The criterion included: QTcF >450 - <=480 mesc, >480 - <=500 msec, >500 msec, increase from baseline >30 - <=60 msec and increase from baseline >60 msec. QT interval >450 - <=480 msec, >480 - <=500 msec, >500 msec, increase from baseline >30 - <=60 msec and increase from baseline >60 msec. Heart rate increase from baseline >25% and value >100 bpm and decrease from baseline >25% and value <60 bpm. PR interval increase from baseline >25% and value >200 msec. QRS interval increase from baseline >25% and value >110 msec. Any new post-baseline notable ECG findings in the DDI phase was collected and reported in this outcome measure.
Time Frame: After 1st dose of encorafenib/binimetinib on Day 1 and up to Day 28 visit in the DDI Phase
Population: All participants who received at least 1 dose of encorafenib/binimetinib. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Number; unit: Count of Participants
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion | Arm 3 - Modafinil
Number analyzed (Participants) | 27 | 12 | 15
Count of Participants
  New QTcF >450 - <=480 mesc: number analyzed (Participants) | 23 | 11 | 13
  New QTcF >450 - <=480 mesc | 6 | 3 | 2
  New QTcF >480 - <=500 msec: number analyzed (Participants) | 27 | 11 | 14
  New QTcF >480 - <=500 msec | 1 | 0 | 1
  New QTcF >500 msec | 0 | 1 | 0
  New QTcF Increase from baseline >30 - <=60 msec | 5 | 3 | 2
  New QTcF Increase from baseline >60 msec | 0 | 0 | 0
  New QT >450 - <=480 msec: number analyzed (Participants) | 26 | 10 | 14
  New QT >450 - <=480 msec | 6 | 0 | 4
  New QT >480 - <=500 msec: number analyzed (Participants) | 27 | 12 | 14
  New QT >480 - <=500 msec | 1 | 1 | 1
  New QT >500 msec: number analyzed (Participants) | 27 | 12 | 14
  New QT >500 msec | 0 | 0 | 0
  New QT Increase from baseline >30 - <=60 msec | 13 | 5 | 9
  New QT Increase from baseline >60 msec | 2 | 0 | 1
  New Heart rate Increase from baseline >25% and value >100 bpm | 0 | 0 | 0
  New Heart rate Decrease from baseline >25% and value <60 bpm | 0 | 0 | 0
  New PR Increase from baseline >25% and value >200 msec: number analyzed (Participants) | 26 | 12 | 15
  New PR Increase from baseline >25% and value >200 msec | 2 | 1 | 3
  New QRS Increase from baseline >25% and value >110 msec | 0 | 1 | 0

148. Secondary Outcome: Number of Participants With Left Ventricular Ejection Fraction (LVEF) Abnormalities in the DDI Phase
Description: LVEF abnormalities are defined according to CTCAE grade version 4.03. Participants was considered as having a LVEF abnormality if the worst post-baseline value was Grade 2, 3, or 4 according to the following classification: Grade 0: Non-missing value below Grade 2; Grade 2: LVEF between 40% and 50% or absolute change from baseline between -10% and <-20%; Grade 3: LVEF between 20% and 39% or absolute change from baseline lower than or equal to -20%; Grade 4: LVEF lower than 20%.
Time Frame: After 1st dose of encorafenib/binimetinib on Day 1 and up to Day 28 visit in the DDI Phase
Population: All participants who received at least 1 dose of encorafenib/binimetinib.
Measure: Number; unit: Count of Participants
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion | Arm 3 - Modafinil
Number analyzed (Participants) | 27 | 12 | 15
Count of Participants | 4 | 2 | 0

149. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Post-DDI Phase
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were those with initial onset or increasing in severity between the first dose of encorafenib/binimetinib and up to 30 days after treatment discontinuation. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. SAEs were adjudicated according to the investigator's assessment. Treatment-related AEs and SAEs were determined by the investigator. Any significant findings in the laboratory test, physical examinations, ophthalmic examinations, vital signs, ECG tests were captured as an AE.
Time Frame: After 1st dose of encorafenib/binimetinib on Day 1 up to 30 days after the post-DDI Phase
Population: All participants who received at least 1 dose of encorafenib/binimetinib.
Measure: Number; unit: Count of Participants
Arm/Group | Arm 1 - CYP Probe Cocktail | Arm 2 - Rosuvastatin and Bupropion | Arm 3 - Modafinil
Number analyzed (Participants) | 25 | 12 | 15
Count of Participants
  Participants with all-causality TEAEs | 17 | 5 | 4
  Participants with treatment-related TEAEs | 10 | 2 | 2
  Participants with all-causality SAEs | 11 | 3 | 4
  Participants with treatment-related SAEs | 4 | 0 | 1
  AEs leading to study drug discontinuation (all-causality) | 4 | 1 | 2
  AEs leading to study drug discontinuation (treatment-related) | 2 | 0 | 1
  AEs requiring dose interruption (all-causality) | 10 | 3 | 1
  AEs requiring dose interruption (treatment-related) | 7 | 2 | 1
  AEs requiring dose reduction (all-causality) | 1 | 0 | 0
  AEs requiring dose reduction (treatment-related) | 1 | 0 | 0
  AEs requiring additional therapy (all-causality) | 14 | 4 | 2
  AEs requiring additional therapy (treatment-related) | 7 | 2 | 0
  Deaths | 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: DDI phase was the period after the 1st dose of encorafenib-binimetinib on Day 1 and up to Day 28 visit for Arm 1, Arm 2 and Arm 3. Post-DDI phase was the period after the 1st dose of encorafenib-binimetinib on Day 1 up to 167.0 weeks for Arm 1, up to 48.1 weeks for Arm 2 and 67.9 weeks for Arm 3
Description: An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both serious and non-serious event. Safety population included all participants who received at least one dose of encorafenib and/or binimetinib.
Groups:
- Arm 1 - CYP Probe Cocktail (DDI Phase); Arm 1 - CYP Probe Cocktail （Post-DDI Phase): Participants received a single oral dose of the CYP probe cocktail (losartan tablet 25 mg, dextromethorphan capsule 30 mg, caffeine liquid 50 mg, omeprazole capsule 20 mg, and midazolam syrup 2 mg) on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
- Arm 2 - Rosuvastatin and Bupropion (DDI Phase); Arm 2 - Rosuvastatin and Bupropion (Post-DDI Phase): Participants received a single oral dose of rosuvastatin tablet 10 mg and bupropion IR tablet 75 mg on Day -7, Day 1, and Day 14. Encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) were continuously administered initiated on Day 1 until treatment discontinuation criteria were met. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 35 days (Day -7 to Day 28).
- Arm 3 - Modafinil (DDI Phase); Arm 3 - Modafinil (Post-DDI Phase): Participants received continuous treatment with encorafenib (capsule, 450 mg QD) and binimetinib (tablet, 45 mg BID) from Day 1 until treatment discontinuation criteria were met. Continuous treatment of modafinil (tablet, 400 mg QD) was started on Day 15 through Day 21. All study interventions were taken within 10 minutes. There were 2 treatment phases, a DDI phase followed by a post-DDI phase. The duration of the DDI phase was 28 days (Day 1 to Day 28).
Arm/Group | Arm 1 - CYP Probe Cocktail (DDI Phase) | Arm 2 - Rosuvastatin and Bupropion (DDI Phase) | Arm 3 - Modafinil (DDI Phase) | Arm 1 - CYP Probe Cocktail （Post-DDI Phase) | Arm 2 - Rosuvastatin and Bupropion (Post-DDI Phase) | Arm 3 - Modafinil (Post-DDI Phase)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/12 | 0/15 | 1/25 | 2/12 | 3/15
Serious Adverse Events (participants affected / at risk) | 2/27 | 1/12 | 0/15 | 11/25 | 3/12 | 4/15
Other Adverse Events (participants affected / at risk) | 25/27 | 9/12 | 11/15 | 4/25 | 4/12 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - CYP Probe Cocktail (DDI Phase) (N=27) | Arm 2 - Rosuvastatin and Bupropion (DDI Phase) (N=12) | Arm 3 - Modafinil (DDI Phase) (N=15) | Arm 1 - CYP Probe Cocktail （Post-DDI Phase) (N=25) | Arm 2 - Rosuvastatin and Bupropion (Post-DDI Phase) (N=12) | Arm 3 - Modafinil (Post-DDI Phase) (N=15)
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 2
Pyrexia (General disorders) | 2 | 1 | 0 | 2 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - CYP Probe Cocktail (DDI Phase) (N=27) | Arm 2 - Rosuvastatin and Bupropion (DDI Phase) (N=12) | Arm 3 - Modafinil (DDI Phase) (N=15) | Arm 1 - CYP Probe Cocktail （Post-DDI Phase) (N=25) | Arm 2 - Rosuvastatin and Bupropion (Post-DDI Phase) (N=12) | Arm 3 - Modafinil (Post-DDI Phase) (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 1 | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
Periorbital discomfort (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Serous retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 5 | 4 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 3 | 4 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 3 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 2 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 3 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 3 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 6 | 0 | 2 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Optic disc drusen (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 6 | 0 | 0 | 2 | 0 | 0
Amylase increased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT03864042/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT03864042/SAP_001.pdf